CLINICAL TRIAL: NCT04968808
Title: OPtimal TIming of Fractional Flow Reserve-Guided Complete RevascularizatiON in Non-ST-Segment Elevation Myocardial Infarction (OPTION-NSTEMI)
Brief Title: Timing of FFR-guided PCI for Non-IRA in NSTEMI and MVD (OPTION-NSTEMI)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chonnam National University Hospital (Other)
Responsible Party: Principal Investigator, Min Chul Kim, Associate Professor, Chonnam National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CNUH-2021-223
Record Dates: First submitted 2021-07-09; First posted 2021-07-20 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-02

CONDITIONS: Myocardial Infarction, Acute; Multi-Vessel Coronary Artery Stenosis; Multi Vessel Coronary Artery Disease
Keywords: Non-ST-Segment Elevation Myocardial Infarction; Multi-Vessel Coronary Artery Disease; Multi-Vessel Coronary Artery Stenosis; Culprit-Only; Multi-Vessel Percutaneous Coronary Intervention; Percutaneous Coronary Intervention; Complete Revascularization; Timing; Staged Percutaneous Coronary Intervention; Fractional Flow Reserve
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Staged in-hospital CR (complete revascularization) (Active Comparator): Non-infarct related artery (IRA) will be revascularized in other day (during hospitalization) after percutaneous coronary intervention (PCI) for IRA. Non-IRA lesion which have equal or more than 70% diameter stenosis by visual estimation will be revascularized without fractional flow reserve (FFR) evaluation. Non-IRA lesion with diameter stenosis 50-69% by visual estimation will be evaluated using FFR device. In case of FFR value more than 0.8, non-IRA lesion wll be deferred without PCI. If FFR value was equal or less than 0.8, non-IRA lesion will be revascularized.
  Interventions: Procedure: Staged in-hospital complete revascularization
- Immediate CR (complete revascularization) (Experimental): Non-infarct related artery (IRA) will be revascularized immediately after percutaneous coronary intervention (PCI) for IRA (during index PCI). Non-IRA lesion which have equal or more than 70% diameter stenosis by visual estimation will be revascularized without fractional flow reserve (FFR) evaluation. Non-IRA lesion with diameter stenosis 50-69% by visual estimation will be evaluated using FFR device. In case of FFR value more than 0.8, non-IRA lesion wll be deferred without PCI. If FFR value was equal or less than 0.8, non-IRA lesion will be revascularized.
  Interventions: Procedure: Immediate complete revascularization

INTERVENTIONS:
Procedure: Staged in-hospital complete revascularization — Patients with non-ST-segment elevation myocardial infarction and multivessel disease will be randomized after percutaneous coronary intervention (PCI) for infarct-related artery (IRA). All patients will be randomized to immediate complete revascularization group or staged revascularization group by 1:1 fashion. Staged in-hospital complete revascularization group will receive staged PCI for non-IRA in other day (during hospitalization) after PCI for IRA. Non-IRA lesion which have equal or more than 70% diameter stenosis by visual estimation will be revascularized without fractional flow reserve (FFR) evaluation. Non-IRA lesion with diameter stenosis 50-69% by visual estimation will be evaluated using FFR device. In case of FFR value more than 0.8, non-IRA lesion wll be deferred without PCI. If FFR value was equal or less than 0.8, non-IRA lesion will be revascularized.
  Arms: Staged in-hospital CR (complete revascularization)
Procedure: Immediate complete revascularization — Patients with non-ST-segment elevation myocardial infarction and multivessel disease will be randomized after percutaneous coronary intervention (PCI) for infarct-related artery (IRA). All patients will be randomized to immediate complete revascularization group or staged revascularization group by 1:1 fashion. Immediate complete revascularization group will receive simultaneous PCI for both IRA and non-IRA during index PCI. Non-IRA lesion which have equal or more than 70% diameter stenosis by visual estimation will be revascularized without fractional flow reserve (FFR) evaluation. Non-IRA lesion with diameter stenosis 50-69% by visual estimation will be evaluated using FFR device. In case of FFR value more than 0.8, non-IRA lesion wll be deferred without PCI. If FFR value was equal or less than 0.8, non-IRA lesion will be revascularized.
  Arms: Immediate CR (complete revascularization)

SUMMARY:
Many patients with non-ST-segment elevation myocardial infarction (NSTEMI) have multivessel coronary artery disease (MVD), which is associated with poor clinical outcomes. However, there have been few studies regarding revascularization strategy in patients with NSTEMI and MVD. Therefore, we planned to perform prospective, open-label, randomized trial to evaluate the efficacy and safety of immediate complete revascularization (percutaneous coronary intervention [PCI] for both infarct-related artery [IRA] and non-IRA during index PCI) compared to staged PCI strategy of non-IRA (PCI for IRA followed by non-IRA PCI after several days). PCI procedure at non-IRA with diameter stenosis between 50 and 69% should be conducted with the aid of fractional flow reserve (FFR), and non-IRA with diameter stenosis ≥ 70% will be revascularized without FFR.

DETAILED DESCRIPTION:
Many patients with non-ST-segment elevation myocardial infarction (NSTEMI) have multivessel coronary artery disease (MVD), which is associated with poor clinical outcomes. In cases of hemodynamically stable ST-segment elevation myocardial infarction (STEMI) and MVD, many studies demonstrated the superiority of complete revascularization (CR) by both one-stage and multistage procedures compared to culprit-only revascularization (COR). The 2017 European Society of Cardiology (ESC) guidelines for STEMI recommend routine revascularization for non infarct-related artery (IRA) lesions before hospital discharge in patients without cardiogenic shock.

However, there have been few studies regarding revascularization strategy in patients with NSTEMI and MVD. Only one randomized controlled trial, the SMILE trial (J Am Coll Cardiol 2016;67:264-72), compared one-stage and multi-stage multivessel revascularization (MVR) in these patients. Although the results of most studies analyzing interventional strategies in patients with NSTEMI and MVD showed superior results of MVR compared to COR, they did not provide information about staged revascularization. One-stage MVR was associated with better clinical outcomes compared to multi-stage MVR in the SMILE trial, while one-stage and multi-stage MVR had similar incidences of adverse outcomes in large registry data. Although the 2018 ESC/European Association for Cardio-Thoracic Surgery (EACTS) guidelines for myocardial revascularization recommend complete one-stage revascularization in NSTEMI and MVD, it emphasizes individualization based on clinical status and comorbidities, as well as disease severity. In 2020 ESC guidelines for non-ST-segment elevation acute coronary syndrome, this strategy is maintained. CR during index percutaneous coronary intervention (PCI) is recommended in NSTEMI patients with MVD (class IIb, level B).

Whether to revascularize non-IRA using angiography or fractional flow reserve (FFR) is also problematic. FFR is a useful tool for assessing hemodynamic significance of non-IRA during both acute and subacute stage, and FFR-guided PCI for non-IRA lesion is recommended during index PCI (class IIb, level B). In the SMILE trial, a 25.8% of study patients received FFR-guided PCI for non-IRA. Although FFR is a well-known tool to evaluate significant ischemia of moderate stenosis, the most studies regarding FFR enrolled patients without acute myocardial infarction (AMI).

However, the recommendations in current guidelines, which recommends CR during index PCI, is not sufficiently powered to assess differences in clinical outcomes between interventional strategy. There are also few studies regarding this issue, and discrepancy in clinical outcomes between randomized trial and observational studies. Furthermore, FFR-guided PCI for non-IRA is not mandatory in these studies.

Therefore, we planned to perform prospective, open-label, randomized trial to evaluate the efficacy and safety of immediate complete revascularization (PCI for both IRA and non-IRA during index PCI) compared to staged PCI strategy of non-IRA (PCI for IRA followed by non-IRA PCI after several days). PCI procedure at non-IRA with diameter stenosis between 50 and 69% should be conducted with the aid of FFR, and non-IRA with diameter stenosis ≥ 70% will be revascularized without FFR.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 19 years old
2. Non-ST-segment elevation myocardial infarction

   * Angina pectoris or equivalent ischemic chest discomfort with at least 1 of 3 features and,

     * occurs at rest, usually lasting > 10 minutes
     * severe and new onset (within the prior 4-6 weeks)
     * crescendo pattern
   * Elevated cardiac biomarkers and,

     * ≥ 99% value of high-sensitivity cardiac troponin
   * No ST-segment elevation ≥ 0.1 mV in ≥ 2 contiguous leads or newly developed left bundle branch block on 12-lead electrocardiogram
3. PCI within 72 hours after symptom development
4. Multivessel disease: Non-IRA with at least 2.5 mm diameter and 50% diameter stenosis by visual estimation
5. Patient's or protector's agreement about study design and the risk of PCI

Exclusion Criteria:

1. Cardiogenic shock at initial presentation or after treatment of IRA
2. TIMI flow at non-IRA ≤ 2
3. Severe procedural complications (e.g. persistent no-reflow phenomenon, coronary artery perforation) which restricts study enrollment by operators' decision
4. Non-IRA lesion not suitable for PCI treatment by operators' decision
5. Chronic total occlusion at non-IRA
6. History of anaphylaxis to contrast agent
7. Pregnancy and lactation
8. Life expectancy < 1-year
9. Severe valvular disease
10. History of CABG, or planned CABG
11. Fibrinolysis before admission

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1014 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence rate of all-cause death, non-fatal myocardial infarction, or all unplanned revascularization | Up to 12 months
  Composite endpoint of all-cause death, non-fatal myocardial infarction, or all unplanned revascularization at 1 year from baseline

SECONDARY OUTCOMES:
Rate of contrast-induced nephropathy | Up to 12 months
  Rate of contrast-induced nephropathy during initial hospitalization
Cumulative incidence rate of all unplanned revascularization | Up to 12 months
  Cumulative incidence rate of all unplanned revascularization at each visit
Cumulative incidence rate of target-lesion revascularization | Up to 12 months
  Cumulative incidence rate of target-lesion revascularization at each visit
Cumulative incidence rate of target-vessel revascularization | Up to 12 months
  Cumulative incidence rate of target-vessel revascularization at each visit
Cumulative incidence rate of non-target vessel revascularization | Up to 12 months
  Cumulative incidence rate of non-target vessel revascularization at each visit
Cumulative incidence rate of all-cause death | Up to 12 months
  Cumulative incidence rate of all-cause death at each visit
Cumulative incidence rate of cardiac death | Up to 12 months
  Cumulative incidence rate of cardiac death at each visit
Cumulative incidence rate of non-cardiac death | Up to 12 months
  Cumulative incidence rate of non-cardiac death at each visit
Cumulative incidence rate of non-fatal myocardial infarction | Up to 12 months
  Cumulative incidence rate of non-fatal myocardial infarction at each visit
Cumulative incidence rate of hospitalization for unstable angina | Up to 12 months
  Cumulative incidence rate of hospitalization for unstable angina at each visit
Cumulative incidence rate of hospitalization for heart failure | Up to 12 months
  Cumulative incidence rate of hospitalization for heart failure at each visit
Cumulative incidence rate of definite or probable stent thrombosis | Up to 12 months
  Cumulative incidence rate of definite or probable stent thrombosis at each visit
Cumulative incidence rate of ischemic and hemorrhagic stroke | Up to 12 months
  Cumulative incidence rate of ischemic and hemorrhagic stroke at each visit
Cumulative incidence rate of major bleeding (BARC [Bleeding Academic Research Consortium] definitions type 3 or 5) | Up to 12 months
  Cumulative incidence rate of major bleeding (BARC [Bleeding Academic Research Consortium] definitions type 3 or 5) at each visit

CONTACTS AND LOCATIONS:
Overall Officials: Min Chul Kim, MD, Principal Investigator — Chonnam National University Hospital
Locations (1):
- Chonnam National University Hospital, Gwangju, South Korea

IPD SHARING:
Plan to Share IPD: No